CLINICAL TRIAL: NCT03485170
Title: PET Imaging of Hemophilic Arthropathy Correlates With Clinical, Radiographic and Sonographic Assessments
Brief Title: PET Imaging of Hemophilic Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tsung-Ying Li, Attending Physician, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2-106-05-028
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Hemophilia; Arthropathy; Inflammation
Keywords: Hemophilia; Hemophilic arthropathy; PET
MeSH Terms: conditions — Hemophilia A; Joint Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET (Other): Hemophilia patients receive PET evaluation
  Interventions: Diagnostic Test: 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT — glucose analogue fluorine-18-fluorodeoxyglucose positron emission tomography with computed tomography scan

SUMMARY:
Repeated hemarthroses in patients with hemophilia may lead to hemophilic arthropathy with marked inflammation and synovial hypertrophy. Power Doppler ultrasonography is a useful tool in hemophilic arthropathy for assessment of disease activity and for monitoring response to treatment. Imaging inflammation with glucose analogue fluorine-18-fluorodeoxyglucose positron emission tomography (18F-FDG PET) is based on that infiltrated granulocytes and tissue macrophages use glucose as an energy source. Metabolism and 18F-FDG uptake increase when inflammation occurring. The purpose of this study is to investigate the associations between 18F-FDG PET/CT and Power Doppler assessment in patients with hemophilic arthropathy.

DETAILED DESCRIPTION:
The study will be performed at the Hemophilia Care and Research Center. We will recruit 20 participants. Inclusion criteria included age 20 years and above hemophilia A or B patients who reported history of hemarthroses of knee, ankle, elbow, shoulder or hip joints. Participants will be excluded for any of the following: presence of joint infections, any surgery on the joints in preceding 6 months, history of rheumatoid arthritis or other inflammatory arthropathy, history of major trauma or presence of neoplasm around joints.

We will collect clinically relevant information including age, body mass index (BMI), hemophilia type and severity, inhibitor titre, schedule of prophylaxis therapy with coagulation factor VIII or IX concentrates history of joint hemarthrosis, and bleeding events in the previous one year. The history of joint bleeding and the total number of joint bleeding events in the previous one year will be obtained from medical chart review recorded according to the patient's bleeding diaries.

18F-FDG PET /CT PET/CT will be performed using a Biograph PET/CT scanner (Discovery 710, GE Healthcare, WI, USA). All patients will fast except for water at least 6 hours prior to the examination. Sixty minutes after the intravenous injection of 10 mCi 18F-FDG, imaging will be performed using a spiral CT scan from the shoulder to the ankle with a 5 mm thickness per slice. Subsequently, PET data will be acquired in a supine position. The images will be reviewed by an experienced nuclear medicine physician unaware of the severity of hemophilic arthropathy in USG and plain x-ray. The analysis method is semi-quantitative and applied maximal standardized uptake (SUVmax) values. The SUVmax for each joint will be measured by placing regions of interest (ROIs) on the axial image of the joint. The SUVmax will be calculated as the maximum FDG uptake within the ROI divided by the injected dose over the patient's body weight (SUVmax = maximum pixel activity/[injected dose/body weight]).

Ultrasonography The USG assessment will be performed according to a standard technique using Terason t3000 machines (Teratech™ , Burlington, Massachusetts, USA) with a 5-12 MHz linear transducer. The probe scans the joint in the longitudinal view with the elbow in 90 degree flexion, or the knee or ankle in full extension. Synovium thickness and hyperemia were evaluated from the lateral, middle, and medial aspects of the anterior suprapatellar recess. Power Doppler assessment of selected synovial sites is carried out with settings standardized to a pulse repetition frequency of 700 Hz. The power Doppler gain is adjusted to a level just below the disappearance of artifacts under the bony cortex. The intensity of the blood flow in the synovium is scored into 0 to 3 (0=No flag; 1 = 1 flag; 2 = 2-3 flags; 3=>3 flags) adapted from Klukowska and Melchiorre et al. Averages of synovium thickness and score of hyperemia in lateral, middle, and medial aspects of the joint will be calculated.

Radiological evaluation Anteroposterior and lateral plain radiographs of joints will be performed and scored according to Pettersson classification by the responsible orthopaedic specialist in our hemophilia center. The Pettersson score ranges from 0 to 13 and is based on the following radiographic features of joints: osteoporosis, osteophytes, narrowing of joint space, subchondral irregularity, subchondral cyst formation, erosion of joint margins, and bone remodelling. A totally normal joint has a score of zero. The Pettersson scoring system has been adopted by the World Federation of Hemophilia as the preferred radiographic classification system for hemophilic arthropathy.

Assessment of joint function ROM of joint is measured in degrees with a goniometer according to the American Academy of Orthopedic Surgeons guidelines. All ROM measurements will be performed by the same assessor. The pain intensity will be evaluated subjectively on a visual analogue scale.

For continuous data, the Student's t-test will be used if the data had a normal distribution. The Mann-Witney U test will be performed if a normal distribution was absent. For categorical data, the Chi-square test or Fisher's exact test will be used. The Spearman correlation coefficient will be calculated for each alteration. P value of less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years and above hemophilia A or B patients who reported history of hemarthroses of knee, ankle, elbow, shoulder or hip joints.

Exclusion Criteria:

* resence of joint infections, any surgery on the joints in preceding 6 months, history of rheumatoid arthritis or other inflammatory arthropathy, history of major trauma or presence of neoplasm around joints.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
SUVmax | 1 day
  The analysis method is semi-quantitative and applied maximal standardized uptake (SUVmax) values. The SUVmax for each joint will be measured by placing regions of interest (ROIs) on the axial image of the joint. The SUVmax will be calculated as the maximum FDG uptake within the ROI divided by the injected dose over the patient's body weight (SUVmax = maximum pixel activity/[injected dose/body weight]).

SECONDARY OUTCOMES:
Hyperemia | 1 day
  Power Doppler assessment of selected synovial sites is carried out with settings standardized to a pulse repetition frequency of 700 Hz. The power Doppler gain is adjusted to a level just below the disappearance of artifacts under the bony cortex (9, 13). The intensity of the blood flow in the synovium is scored into 0 to 3 (0=No flag; 1 = 1 flag; 2 = 2-3 flags; 3=>3 flags) adapted from Klukowska and Melchiorre et al
Pettersson score | 1 day
  The Pettersson score ranges from 0 to 13 and is based on the following radiographic features of joints: osteoporosis, osteophytes, narrowing of joint space, subchondral irregularity, subchondral cyst formation, erosion of joint margins, and bone remodelling. A totally normal joint has a score of zero.
ROM of joints | 1 day
  ROM of joint is measured in degrees with a goniometer. Shoulder:0-180; Elbow:0-150; Hip:0-120; Knee:0-135; Ankle:0-70
Pain | 1 day
  The pain intensity will be evaluated subjectively on a visual analogue scale,0(no pain)-10cm(severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Hemophilia care and research center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No